CLINICAL TRIAL: NCT00827151
Title: "2008P-00346: Bone Mass Accrual in Adolescent Athletes"
Brief Title: Bone Mass Accrual in Adolescent Athletes
Acronym: 838
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was not funded
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Madhusmita Misra, Professor Pediatrics, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008P00246; NIH-HCNRC
Record Dates: First submitted 2009-01-16; First posted 2009-01-22 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Amenorrhea; Bone Loss
Keywords: amenorrhea; athletes; bone loss; eumenorrhea
MeSH Terms: conditions — Amenorrhea; Bone Diseases, Metabolic | interventions — Estrogens; Estradiol; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Estrogen and lifestyle (Active Comparator)
  Interventions: Drug: Estrogen
- Lifestyle (No Intervention)

INTERVENTIONS:
Drug: Estrogen — Estrogen 100 mcg patch twice weekly with 10 days of oral progesterone monthly for 12 months versus no medication
  Other Names: Vivelle-Dot; Prometrium
  Arms: Estrogen and lifestyle

SUMMARY:
The adolescent and young adult years are a critical window in time for bone mineral accrual. More than 90% of peak bone mass is achieved by 18 years, and data indicate that insults sustained during adolescence and young adulthood may result in permanent deficits in bone accrual. Adult athletes with amenorrhea (AA) have low bone mineral density (BMD) secondary to hypogonadism, associated with increased fracture risk and associated co-morbidities. We will examine whether estrogen replacement will increase BMD and improve measures of bone microarchitecture in adolescents and young women with AA, thus optimizing peak bone mass.

DETAILED DESCRIPTION:
Young female athletes 18-21 years old will be randomized to estrogen (and progesterone) with lifestyle modification versus lifestyle modification alone for a 12 month period. Bone density and structure will be assessed over this period. Hormonal evaluations will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-21 years of age
* Hypothalamic amenorrhea
* Greater than or equal to 15 years bone age
* BMI between 10th-90th percentiles for age

Exclusion Criteria:

* Use of medications affecting bone metabolism including estrogen/ progesterone, anabolic steroids and glucocorticoids except local application of glucocorticoid creams (washout period of three months necessary prior to study enrollment if medically permissible to discontinue these)
* Presence of anorexia nervosa or %IBW of < 85% based on the 50th %ile of BMI for age
* Spine BMD Z-score < -3
* Conditions other than endurance training that may cause amenorrhea including PCOS (clinical or preceding laboratory evidence of hyperandrogenism with amenorrhea)
* Conditions other than endurance training that may cause bone metabolism to be affected
* Abnormal TSH, elevated FSH, hematocrit < 30%
* Pregnancy

For girls with AA (to be randomized to estrogen and progesterone or no treatment)

* History of migraines, hypertension, allergy to peanut oil, undiagnosed abnormal genital bleeding, known, suspected or history of breast or genital cancer or estrogen dependent neoplasia, known hypersensitivity to progesterone or estrogen or other product ingredients, liver dysfunction or disease
* LFTs greater than 1.5 times the upper limit of normal
* Family history or personal history of conditions that may increase risk of thromboembolism:

  1. Family history of myocardial infarction or strokes occurring at less than 50 years
  2. Family history of clotting disorders: normal coagulation profile will be necessary for enrollment
* History of smoking >10 cigarettes a day (history of smoking >14 cigarettes a day is a contraindication for estrogen, but we will be more conservative in our exclusion criteria)
* Personal history of blood clots

Ages: 18 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2011-05 (Actual); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Bone density | One year

CONTACTS AND LOCATIONS:
Overall Officials: Madhu Misra, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States